CLINICAL TRIAL: NCT02632474
Title: ART Drug Dosage Adjustment Using FSCII in Chinese HIV-infected Population
Brief Title: ART Drug Dosage Adjustment in HIV-infected Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Hongzhou Lu, Doctor, Shanghai Public Health Clinical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FSCII-ART-1
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: HIV Infections
Keywords: HIV Infections; Tenofovir; Efavirenz
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low-dose (Experimental): Tenofovir(TDF)+Lamivudine(3TC)+Efavirenz(EFV)
  Interventions: Drug: Tenofovir(TDF)+Lamivudine(3TC)+Efavirenz(EFV)

INTERVENTIONS:
Drug: Tenofovir(TDF)+Lamivudine(3TC)+Efavirenz(EFV) — The first 2 weeks, TDF (300 mg) + 3-TC (300 mg) + EFV (400 mg); week 3, TDF (200 mg) + 3-TC (300 mg) + EFV (400 mg ); week 4, TDF (150 mg) + 3-TC (300 mg) + EFV (400 mg).From week5, if the HIV viral load decreased as expected or no rebound, use TDF (200 mg) + 3-TC (300 mg) + EFV (400 mg) until study complete; if the viral load increases, switch to the standard treatment regimen: TDF (300 mg) + 3-TC (300 mg) + EFV (600 mg).

SUMMARY:
The purpose of this study is to determine efficacy of the combination of low dose of Tenofovir, Efavirenz and Lamivudine in treating HIV-infection.

DETAILED DESCRIPTION:
The feedback system control (FSC) technique has been developed to rapidly identify optimal combinations for therapeutic purposes. Low dose of TDF+3TC+EFV combination has been test in vitro study by FSC which showed high efficacy and now the investigators apply it to human to further optimize the ART combination.

ELIGIBILITY:
Inclusion Criteria:

* HIV antibody positive
* HIV RNA below 10*E5 copies/ml
* CD4 T cell count above 200 cells/ml
* Provision of written informed consent

Exclusion Criteria:

* HIV genotyping resistant to investigating drug
* Pregnant, breastfeeding, or lactating
* Any serious or active medical or psychiatric illness which, in the opinion of the Investigator, would interfere with treatment, assessment, compliance with the protocol, or subject safety. This would include any active clinically significant renal, cardiac, pulmonary, vascular, or metabolic (thyroid disorders, adrenal disease) illness, or malignancy
* Medical or psychiatric condition or occupational responsibilities that may preclude compliance with the protocol
* Laboratory blood values:
* Haemoglobin <7.0 grams/decilitre (g/dL)
* Neutrophil count <500/mm3
* Platelet count <50,000/mm3
* Aspartate aminotransferase or Alanine transaminase >5 times Upper Limit of Normal (ULN)
* Subjects with an estimated creatinine clearance of <50 mL/minute

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HIV viral load | 48 weeks

SECONDARY OUTCOMES:
CD4 Count | 48 weeks

OTHER OUTCOMES:
Drug Plasma Concentration | Day 7,14,21,28

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China